CLINICAL TRIAL: NCT00439270
Title: Phase I/II Study of Dasatinib and Docetaxel in Metastatic Hormone Refractory Prostate Cancer
Brief Title: Study of Dasatinib and Docetaxel in Metastatic Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-086
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Results first posted 2013-11-27 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Metastatic Prostate Cancer
Keywords: Metastatic hormone refractory prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dasatinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dasatinib, 50 mg + Docetaxel, 60 mg/m^2 (Active Comparator): Participants received dasatinib, 50 mg, administered orally once daily. Docetaxel was administered every 3 weeks as an infusion at 60 mg/m^2.
  Interventions: Drug: Dasatinib; Drug: Docetaxel
- Dasatinib, 50 mg + Doxetaxel, 75 mg/m^2 (Active Comparator): Participants received dasatinib, 50 mg administered orally once daily. Docetaxel was administered every 3 weeks as an infusion at 75 mg/m^2.
  Interventions: Drug: Dasatinib; Drug: Docetaxel
- Dasatinib, 70 mg + Docetaxel, 75 mg/m^2 (Active Comparator): Participants received dasatinib, 70 mg, administered orally once daily. Docetaxel was administered every 3 weeks as an infusion at 75 mg/m^2.
  Interventions: Drug: Dasatinib; Drug: Docetaxel
- Dasatinib, 100 mg + Docetaxel, 75 mg/m^2 (Active Comparator): Participants received dasatinib, 100 mg, administered orally once daily. Docetaxel was administered every 3 weeks as an infusion at 75 mg/m^2.
  Interventions: Drug: Dasatinib; Drug: Docetaxel
- Dasatinib, 120 mg + Docetaxel, 75 mg/m^2 (Active Comparator): Participants received dasatinib, 120 mg, administered orally once daily. Docetaxel was administered every 3 weeks as an infusion at 75 mg/m^2.
  Interventions: Drug: Dasatinib; Drug: Docetaxel

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 50, 70, 100, or 120 mg once daily; treatment may continue until disease progression
  Other Names: Sprycel; BMS-354825
Drug: Docetaxel — Infusion, 60 or 75 mg/m^2, administered every 3 weeks.

SUMMARY:
The purpose of this study is to find the recommended doses of dasatinib and docetaxel given in combination to men with metastatic hormone refractory prostate cancer and to assess the pharmacokinetic interactions between the 2 drugs.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate that was clinically refractory to hormone therapy
* Eastern Cooperative Oncology Group performance status of 0 - 2
* Evidence of progressive metastatic disease at time of enrollment
* Measurable disease on either computer tomography scan or magnetic resonance imaging or positive bone scan with any level of serum prostate specific antigen (PSA) ≥5 ng/ml. Patients with PSA ≥5 ng/ml only and no other radiographic evidence of metastatic prostate cancer were not eligible
* Evidence of progressive disease since the most recent change in therapy. Progressive disease was defined as any one of the following:

  * Objective disease progression: Objective evidence of increase in radiographic lesions or the appearance of 1 or more new lesions
  * Bone scan progression: Appearance of either of the following: 2 or more new lesions on bone scan attributable to prostate cancer or 1 new lesion on bone scan attributable to prostate cancer in conjunction with a rising PSA
  * PSA progression: 2 consecutively rising PSA levels (≥5 ng/mL) separated by 2 weeks with a testosterone concentration of ≤50 ng/dL at 2 week intervals
* Serum testosterone levels ≤50 ng/dL, determined within 2 weeks prior to starting treatment
* Maintaining castrate status: patients who had not undergone surgical orchiectomy must have continued on medical therapies, such as gonadotropin-releasing hormone analogs, to maintain castrate levels of serum testosterone. Those receiving an antiandrogen as part of their first-line hormonal therapy must have shown progression of disease off of the antiandrogen prior to enrollment (6 weeks withdrawal for bicalutamide; 4 weeks for flutamide)

Key Exclusion Criteria:

* Sexually active fertile men not using effective birth control if their partners were women of child-bearing potential
* Known brain metastases
* Clinically-significant cardiovascular disease, including myocardial infarction or ventricular tachyarrhythmia within 6 months; prolonged heart rate-corrected QT interval (QTc) >450 msec; ejection fraction <40%, or major conduction abnormality (unless a cardiac pacemaker was present)
* Pleural or pericardial effusion, due to concerns that the combination of docetaxel and dasatinib could worsen these events
* Uncontrolled intercurrent illness including, ongoing or active infection, cardiac arrhythmia, or psychiatric illness/social situations that limit compliance with study requirements
* Participants were permitted to continue on a daily multivitamin but all other herbal, alternative, and food supplements must have been discontinued before enrollment into the study
* Ketoconazole must have been discontinued 4 weeks prior to enrollment
* Patients were not permitted to receive radioactive bone targeting agents, such as Strontium or Samarian ,while on study treatment
* The following restrictions on prior therapy for metastatic disease applied:

  * One chemotherapy regimen was permitted as long as docetaxel resistance or intolerance was not demonstrated. Docetaxel resistance was defined as objective disease progression or confirmed PSA progression during docetaxel therapy or within 3 months of treatment completion. Docetaxel intolerance was defined as toxicity requiring docetaxel interruption >4 weeks or dose modification below approved doses
  * No more than 1 prior course of palliative radiotherapy
  * Up to 1 prior treatment with a nonchemotherapeutic agent was permitted as treatment for metastatic prostate cancer
  * No prior radioisotope therapy with Strontium-89, Samarium, or similar agents
  * No limitation on prior hormonal therapy
  * QTc prolonging agents strongly associated with Torsade de Pointes arrhythmia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-07; Primary Completion 2012-02 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (5):
  - University of Chicago, Chicago, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Hematology-Oncology Associates Of Rockland, Nyack, New York
  - Duke University, Durham, North Carolina
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Araujo JC, Mathew P, Armstrong AJ, Braud EL, Posadas E, Lonberg M, Gallick GE, Trudel GC, Paliwal P, Agrawal S, Logothetis CJ. Dasatinib combined with docetaxel for castration-resistant prostate cancer: results from a phase 1-2 study. Cancer. 2012 Jan 1;118(1):63-71. doi: 10.1002/cncr.26204. Epub 2011 Jul 25. PMID 21976132
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 49 participants were enrolled in the study, and 46 entered the treatment period and received at least 1 dose of dasatinib.
Groups:
- Dasatinib, 50 mg + Docetaxel, 75 mg/m^2: Participants received dasatinib, 50 mg administered orally once daily. Docetaxel was administered every 3 weeks as an infusion at 75 mg/m^2.
Period: Phase 1 (18.1 Months)
Arm/Group | Dasatinib, 50 mg + Docetaxel, 60 mg/m^2 | Dasatinib, 50 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 70 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 120 mg + Docetaxel, 75 mg/m^2
Started | 3 (Participants who received treatment) | 3 (Participants who received treatment) | 3 (Participants who received treatment) | 4 (Participants who received treatment) | 3 (Participants who received treatment)
Completed | 0 (Remained on study) | 0 (Remained on study) | 0 (Remained on study) | 4 (Remained on study) | 0 (Remained on study)
Not Completed | 3 | 3 | 3 | 0 | 3
Not completed — Disease progression | 3 | 2 | 3 | 0 | 3
Not completed — Study drug toxicity | 0 | 1 | 0 | 0 | 0
Period: Phase 2 (51.6 Months)
Arm/Group | Dasatinib, 50 mg + Docetaxel, 60 mg/m^2 | Dasatinib, 50 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 70 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 120 mg + Docetaxel, 75 mg/m^2
Started | 0 | 0 | 0 | 34 (Includes 4 patients who completed Phase 1) | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 34 | 0
Not completed — Disease progression | 0 | 0 | 0 | 18 | 0
Not completed — Poor compliance/noncompliance | 0 | 0 | 0 | 1 | 0
Not completed — Study drug toxicity | 0 | 0 | 0 | 6 | 0
Not completed — Maximum clinical benefit | 0 | 0 | 0 | 3 | 0
Not completed — No longer meets study criteria | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0
Not completed — Adverse event unrelated to study drug | 0 | 0 | 0 | 2 | 0
Not completed — Insurance no longer covered patient care | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients who received at least 1 dose of dasatinib
Groups:
- Dasatinib, 50 mg + Docetaxel, 60 mg/m^2: Participants received dasatinib, 50 mg, administered orally once daily. Docetaxel was administered every 3 weeks as an infusion at 60 mg/m^2. Provided no dose-limiting toxicities occurred, at least 3 participants received treatment in each arm.
- Dasatinib, 50 mg + Docetaxel, 75 mg/m^2: Participants received dasatinib, 50 mg, administered orally once daily. Docetaxel was administered every 3 weeks as an infusion at 75 mg/m^2. Provided no dose-limiting toxicities occurred, at least 3 participants received treatment in each arm.
- Dasatinib, 70 mg + Docetaxel, 75 mg/m^2: Participants received dasatinib, 70 mg, administered orally once daily. Docetaxel was administered every 3 weeks as an infusion at 75 mg/m^2. Provided no dose-limiting toxicities occurred, at least 3 participants received treatment in each arm.
- Dasatinib, 100 mg + Docetaxel, 75 mg/m^2: Participants received dasatinib, 100 mg, administered orally once daily. Docetaxel was administered every 3 weeks as an infusion at 75 mg/m^2. Provided no dose-limiting toxicities occurred, at least 3 participants received treatment in each arm.
- Dasatinib, 120 mg + Docetaxel, 75 mg/m^2: Participants received dasatinib, 120 mg, administered orally once daily. Docetaxel was administered every 3 weeks as an infusion at 75 mg/m^2. Provided no dose-limiting toxicities occurred, at least 3 participants received treatment in each arm.
- Total: Total of all reporting groups
Arm/Group | Dasatinib, 50 mg + Docetaxel, 60 mg/m^2 | Dasatinib, 50 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 70 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 120 mg + Docetaxel, 75 mg/m^2 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 34 | 3 | 46
Age, Customized [Number; unit: Participants]
  <65 years | 0 (3.51) | 1 (5.03) | 1 (11.02) | 19 (8.43) | 2 (13.23) | 23
  >=65 years | 3 | 2 | 2 | 15 | 1 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 34 | 3 | 46
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 0 | 0 | 0 | 4 | 0 | 4
  White | 3 | 3 | 3 | 29 | 3 | 41
  Other | 0 | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic/Latino | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic/Latino | 3 | 3 | 3 | 33 | 3 | 45

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With a Prostate Specific Antigen (PSA) Response
Description: PSA response rate is defined as a decrease of >=50% in PSA levels from baseline, sustained for at least 6 weeks and confirmed by at least 2 measurements
Time Frame: At pretreatment visit, and on Day 1 of Cycles 2 through 12, then every other cycle, where investigator deems appropriate, and at end of treatment (up to 51.6 months)
Population: All patients who received dasatinib, 100 mg + docetaxel, 75 mg/m^2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2
Number analyzed (Participants) | 34
Percentage of participants | 64.7 [46.49 to 80.25]

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Dasatinib Administered With Docetaxel
Description: MTD was defined by dose-limiting toxicity (DLT) criteria. DLT was defined as grade 4 neutropenia causing treatment interruption for >14 days, febrile neutropenia, grade 4 thrombocytopenia, grade 3 thrombocytopenia with a bleeding episode requiring platelet transfusion, nausea and/or vomiting despite medical intervention/prophylaxis causing treatment interruption for >14 days, grade 3-4 asthenia/fatigue, any other grade >=3 nonhematologic toxicity except alopecia or transient arthralgia/myalgia (unless unresponsive to intervention), or interruption of study drug for >14 days due to toxicity. When defined, the MTD would serve as recommended Phase 2 dose of each drug in the combination of oral dasatinib and intravenous docetaxel.
Time Frame: From Day 3 of first 21-day cycle to Cycle 2 , Day 21 (or Study Day 42)
Population: All patients who received at least 1 dose of dasatinib in Phase 1
Measure: Number; unit: mg
Groups:
- All Treated (Phase 1): Participants received dasatinib as 50, 70, 100, or 120 mg administered orally once daily with docetaxel, administered every 3 weeks as an infusion at 60 or 75 mg/m^2. A standard 3+3 design was used, in which 3-6 patients were exposed to a dose level combination. Using a dose escalation scheme, the first 3-6 patients received the lower dose level combination. Escalation to the next dose level combination for another set of 3-6 patients was initiated if no dose-limiting toxicities (DLTs) were observed. If 2 or more DLTs were observed for a dose level combination, the MTD was defined as the previous dose level combination.
Arm/Group | All Treated (Phase 1)
Number analyzed (Participants) | 16
mg | NA — Because no DLT occurred, MTD was not determined. Recommended Phase 2 dasatinib dose based on ongoing studies in chronic myelogenous leukemia and previous study in chronic refractory prostate cancer. Recommended docetaxel dose based on package insert.

3. Secondary Outcome: Duration of Prostate Specific Antigen (PSA) Response
Description: Duration of response is computed for participants with confirmed PSA response. It is measured in months from the time of the first of 2 consecutive measurements meeting the criteria for confirmed PSA response to the date of the first of 3 consecutive measurements that confirm PSA progression, the date of disease progression, or the date of death. Participants who neither progressed (PSA or disease) nor died were censored on the date of their last PSA assessment. PSA response is defined as a decrease of >=50% in PSA levels from baseline, sustained for at least 6 weeks and confirmed by at least 2 measurements. PSA progression is defined as 3 consecutive increases in PSA from baseline or nadir, each measurement at least 1 week apart. The final confirming PSA measurement had to be ≥5ng/mL higher than baseline or nadir and also represent at least a 50% increase from baseline or nadir (ie, the value is ≥1.5*baseline or nadir PSA).
Time Frame: At pretreatment visit, and on Day 1 of Cycles 2 through 12, then every other cycle, where investigator deems appropriate, and at end of treatment
Population: All participants who received dasatinib, 100 mg + docetaxel, 75 mg/m^2 and who had a PSA response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2
Number analyzed (Participants) | 22
Months | 9.5 [7.1 to 25.2]

4. Secondary Outcome: Number of Months of Progression-free Survival (PFS)
Description: PFS defined as time in months from the first dosing date to the date of disease progression or the date of death. Patients who neither progressed nor died were censored on the date of their last on-study prostate specific antigen (PSA) measurement, tumor assessment, or radionuclide bone scan assessment (whichever occurred last). Disease progression defined as either of the following: progression on radionuclide bone scan, death, or at least 2 of the following:
  tumor progression, as defined by modified Response Evaluation Criteria in Solid Tumors; PSA progression; or investigator-defined clinical progression based on physical examination, history, symptoms, and performance status.
Time Frame: Patients with an event: time from first dose to disease progression or death, whichever occurs first. Patients without an event: time to last on-study PSA measurement, tumor assessment, or radionuclide bone scan assessment, whichever occurs last
Population: All patients who received dasatinib, 100 mg + docetaxel, 75 mg/m^2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2
Number analyzed (Participants) | 34
Months | 11.5 [8.8 to 18.9]

5. Secondary Outcome: Percentage of Participants With an Objective Tumor Response by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Objective response rate is defined as the percentage of participants who have achieved best responses of confirmed Complete Response (CR) or Partial Response (PR) where confirmed requires repeat evaluations for a minimum of 4 weeks after the criteria for response are first met. RECIST: CR=disappearance of clinical and radiologic evidence of target lesions; PR=a 30% or greater decrease in the sum of the longest diameter (LD) of all lesions in reference to the baseline sum LD.
Time Frame: Pretreatment visit then every 6 weeks thereafter (up to 51.6 months)
Population: All patients who received dasatinib, 100 mg + docetaxel, 75 mg/m^2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2
Number analyzed (Participants) | 34
Percentage of participants | 44.1 [27.19 to 62.11]

6. Secondary Outcome: Number of Participants by Best On-study Tumor Response by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: RECIST for target lesions: Complete Response (CR)=disappearance of clinical and radiologic evidence of target lesions. Partial Response (PR)=a 30% or greater decrease in the sum of the longest diameter (LD) of all lesions in reference to the baseline sum LD. Stable disease (SD)=neither sufficient increase to qualify for Progressive Disease (PD) nor sufficient shrinkage to qualify for PR.
  PD=a 20% or greater increase in the sum of LD of all target lesions, taking as reference the smallest sum LD recorded at or following baseline; unequivocal progression of nonmeasurable disease/lesions as evaluated by CT scan or MRI (not as evaluated by radionuclide bone scan) and/or new lesions are present.
  To qualify as SD, patients had to exhibit SD for a minimum of 18 weeks. Those with evaluations noted as SD prior to 18 weeks and discontinued were reported as no change.
Time Frame: Pretreatment visit then every 6 weeks thereafter (up to 51.6 months)
Population: All patients who received dasatinib, 100 mg + docetaxel, 75 mg/m^2
Measure: Number; unit: Participants
Arm/Group | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2
Number analyzed (Participants) | 34
Participants
  Complete response | 0
  Partial response | 15
  Stable disease | 1
  No change | 3
  Progressive disease | 2
  Not evaluable | 13

7. Primary Outcome: Recommended Phase 2 Dose of Dasatinib Administered With Docetaxel, 75 mg/m^2
Description: Because no dose-limiting toxicities occurred, the recommended dose of dasatinib used in Phase 2 was based on findings from ongoing studies in chronic myelogenous leukemia and experience from the previous Phase 2 study of single-agent dasatinib in chronic refractory prostate cancer. The recommended Phase 2 dose of docetaxel (75 mg/m^2) was based on the docetaxel package insert.
Time Frame: From Day 3 of first 21-day cycle to Cycle 2 , Day 21 (or Study Day 42)
Population: All patients who received at least 1 dose of dasatinib in Phase 1
Measure: Number; unit: mg
Groups:
- All Treated (Phase 1): Participants received dasatinib as 50, 70, 100, or 120 mg administered orally once daily with docetaxel, administered every 3 weeks as an infusion at 60 or 75 mg/m^2. A standard 3+3 design was used, in which 3-6 patients were exposed to a dose level combination. Using a dose escalation scheme, the first 3-6 patients received the lower dose level combination. Escalation to the next dose level combination for another set of 3-6 patients was initiated if no dose-limiting toxicities (DLTs) were observed. If, for a dose level combination, 2 or more DLTs were observed, the maximum tolerated dose was defined as the previous dose level combination.
Arm/Group | All Treated (Phase 1)
Number analyzed (Participants) | 16
mg | 100

8. Secondary Outcome: Number of Participants by Best On-study Bone Scan Assessment From Baseline
Description: Stable=no new lesions appeared at any 6-week assessment or new pain was not developed in an area that was previously visualized for a minimum of 18 weeks; no change=stable disease prior to 18 weeks and then discontinued treatment; progression=2 or more new areas of focal uptake or new adverse clinical symptoms in an area previously visualized; improved=disappearance of at least 1 lesion, no new lesions appearing since the most recent prior assessment, and new pain not developing in an area that was previously visualized.
Time Frame: From Day 1 of therapy to last bone scan assessment (up to 51.6 months)
Population: All patients who received dasatinib, 100 mg + docetaxel, 75 mg/m^2
Measure: Number; unit: Participants
Arm/Group | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2
Number analyzed (Participants) | 34
Participants
  Improved | 8
  Stable | 17
  No change | 7
  Progression | 1
  Not evaluable | 1

9. Secondary Outcome: Percentage of Participants With Improvement on Bone Scan
Description: Improvement=disappearance of at least 1 lesion, no new lesions appearing since the most recent prior assessment, and new pain not developing in an area that was previously visualized
Time Frame: From Day 1 of therapy to last bone scan assessment (up to 51.6 months)
Population: All patients who received dasatinib, 100 mg + docetaxel, 75 mg/m^2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2
Number analyzed (Participants) | 34
Percentage of participants | 23.5 [10.75 to 41.17]

10. Secondary Outcome: Baseline Scores and Changes in Pain Intensity From Baseline on the Brief Pain Inventory Short Form (BPI-sf) Scores Through Cycle 6
Description: The BPI-sf assessed intensity of pain in the last 24 hours as well as impact of pain on daily functions. Patients rated the severity of their pain at its worst, least, and average in the last 24 hours using an 11-point rating scale with endpoints of no pain (0 points) and pain as bad as you can imagine (11 points). They were asked to rate their present pain and pain at the time they completed the BPI-sf. Using an 11-point rating scale with endpoints of does not interfere (0 points) and completely interferes (11 points), the BPI-sf similarly assessed to what extent pain interfered with mood, walking, general activity, work, relations with others, sleep, and enjoyment of life. The BPI-sf also asked patients to mark the location of their pain on a body drawing and included other questions about pain treatment and the extent of pain relief. The BPI-sf was collected in the Phase 2 portion of the study only. For on-treatment visits, the BPI-sf was completed prior to the docetaxel infusion.
Time Frame: At pretreatment visit and on Day 1 of Cycles 2 through 6, then Day 1 of every other cycle, at end of treatment, and at follow-up visit
Population: All patients who received dasatinib, 100 mg + docetaxel, 75 mg/m^2, in the Phase 2 portion of the study and completed the BPI-sf at baseline. n=evaluable participants in that cycle.
Measure: Median (Full Range); unit: Units on a scale
Groups:
- Dasatinib, 100 mg + Docetaxel, 75 mg/m^2 (Phase 2 ): Participants received dasatinib, 100 mg, administered orally once daily. Docetaxel was administered every 3 weeks as an infusion at 75 mg/m^2.
Arm/Group | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2 (Phase 2 )
Number analyzed (Participants) | 18
Units on a scale
  Baseline: Average of pain (n=18) | 1.0 [1.0 to 5.8]
  Baseline: Average of pain interference (n=18) | 1.0 [0.0 to 7.3]
  Cycle 2: Average of pain (n=11) | -0.8 [-2.3 to 0.8]
  Cycle 2: Average of pain interference (n=11) | 0.0 [-2.3 to 1.0]
  Cycle 3: Average of pain (n=7) | -0.5 [-2.0 to 0.8]
  Cycle 3: Average of pain interference (n=7) | -0.0 [-3.0 to 1.7]
  Cycle 4: Average of pain (n=10) | -1.0 [-1.5 to 0.0]
  Cycle 4: Average of pain interference (n=10) | -0.1 [-1.0 to 1.6]
  Cycle 5: Average of pain (n=5) | -0.8 [-1.5 to 2.5]
  Cycle 5: Average of pain interference (n=5) | 0.0 [-0.6 to 4.6]
  Cycle 6: Average of pain (n=9) | -0.8 [-1.5 to 0.9]
  Cycle 6: Average of pain interference (n=9) | 0.0 [-1.0 to 4.0]

11. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Drug-related SAEs, Drug-related Adverse Events (AEs), Drug-related AEs Leading to Discontinuation, and Drug-related Grade 3 or 4 AEs in the Overall Population
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Drug-related=having certain, probable, possible, or missing relationship to study drug. Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Leading to death.
Time Frame: From first dose Day 1 through at least 30 days after last dose of either dasatinib or docetaxel, whichever was later (up to approximately 49 months)
Population: All participants who received at least 1 dose of dasatinib
Measure: Number; unit: Participants
Groups:
- All Treated: Participants received dasatinib, 50, 70, 100, or 120 mg, administered orally once daily. Docetaxel was administered every 3 weeks as an infusion at 60 or 75 mg/m^2.
Arm/Group | All Treated
Number analyzed (Participants) | 46
Participants
  Deaths | 3
  SAEs | 17
  Drug-related SAEs | 8
  Drug-related AEs | 45
  Drug-related AEs leading to discontinuation | 7
  Drug-related Grade 3 or 4 AEs | 13

12. Secondary Outcome: Number of Participants With Death as Outcome, Drug-related Serious Adverse Events (SAEs), Drug-related Adverse Events (AEs), Drug-related AEs Leading to Discontinuation, and Drug-related Grade 3 or 4 AEs in the Phase 2 Cohort
Description: as for outcome 11
Time Frame: as for outcome 11
Population: All patients who received dasatinib, 100 mg + docetaxel, 75 mg/m^2
Measure: Number; unit: Participants
Arm/Group | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2
Number analyzed (Participants) | 34
Participants
  Deaths | 2
  Drug-related SAEs | 7
  Drug-related AEs | 33
  Drug-related AEs leading to discontinuation | 6
  Drug-related Grade 3 or 4 AEs | 12

13. Secondary Outcome: Area Under the Concentration-time Curve (AUC) From 0 to 10 Hours Postdose (AUC [0-10])and AUC in 1 Dosing Interval, From Time 0 to 24 Hours (AUC[Tau])of Dasatinib Coadministered With Docetaxel
Time Frame: Cycle 1, Day 14 at 0, 0.5 , 1, 2, 3, 4, 7, 10, and 24 hours postdose
Population: All patients who received at least 1 dose of dasatinib; n=number of patients who were evaluable
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Dasatinib, 50 mg + Docetaxel, 60 mg/m^2 | Dasatinib, 50 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 70 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 120 mg + Docetaxel, 75 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 34 | 3
ng.h/mL
  AUC(0-10) (n=3, 1, 3, 28, 3) | 173.13 (54) | 71.75 (NA) — Insufficient participants with events | 149.79 (26) | 277.07 (54) | 461.82 (35)
  AUC(tau) (n=3, 1, 3, 21, 3) | 205.43 (57) | 82.20 (NA) — Insufficient participants with events | 200.63 (25) | 389.66 (48) | 556.47 (36)

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Dasatinib and of Docetaxel
Time Frame: Docetaxel: Cycle 1, Day 1 at 0, 0.5, 1, 1.25, 1.5, 2, 3, 4, 7, 10, 24, and 48 hours postdose; dasatanib: Cycle 1, Day 14 at 0, .5, 1, 2, 3, 4, 7, 10, and 24 hours postdose
Population: All patients who received at least 1 dose of dasatinib; n=number of patients who were evaluable
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dasatinib, 50 mg + Docetaxel, 60 mg/m^2 | Dasatinib, 50 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 70 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 120 mg + Docetaxel, 75 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 34 | 3
ng/mL
  Dasatinib (n=3, 1, 3, 29, 3) | 42.70 (68) | 21.99 (NA) — Insufficient participants with events | 30.00 (17) | 83.91 (74) | 164.99 (26)
  Docetaxel (n=3, 3, 3, 34, 3) | 2226.25 (46) | 1763.34 (25) | 1748.43 (20) | 2125.49 (33) | 2412.41 (14)

15. Secondary Outcome: Area Under the Concentration-time Curve (AUC) From Time 0 to Infinity (AUC[Inf]) of Docetaxel
Time Frame: Cycle 1, Day 1 at 0, 0.5, 1, 1.25, 1.5, 2, 3, 4, 7, 10, 24, and 48 hours postdose
Population: All patients who received at least 1 dose of dasatinib
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Dasatinib, 50 mg + Docetaxel, 60 mg/m^2 | Dasatinib, 50 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 70 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 120 mg + Docetaxel, 75 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 34 | 3
ng.h/mL | 3085.59 (54) | 2064.49 (24) | 2113.37 (23) | 2663.83 (33) | 3283.27 (19)

16. Secondary Outcome: Number of Participants Meeting the Criteria for On-study Abnormal Results Grade 3-4 of Clinical Laboratory Tests
Description: ULN=upper limit of normal. Graded by Common Toxicity Criteria: 1 (least severe) to 4 (life threatening ). Absolute neutrophil count (*10^9/L), Grade 3, <1.0-0.5; Grade 4, <0.5. Hemoglobin (mmol/L), Grade 3, <4.9-4.0; Grade 4, <4.0. Platelets (*10^9/L), Grade 3, <50.0-25.0; Grade 4, <25.0. Leukocytes (*10^9/L) Grade 3, <2.0-1.0; Grade 4, <1.0. ALP, ALT, and AST (*ULN), Grade 3, >5.0-20.0; Grade 4, >20.0. Total bilirubin (*ULN), Grade 3, >3.0-10.0; Grade 4, >10.0. Creatinine (*ULN), Grade 3, >3.0-6.0; Grade 4, >6.0. Hypercalcemia (mmol/L), Grade 3, >3.1-3.4; Grade 4, >3.4. Hypocalcemia mmol/L), Grade 3, <1.75-1.5; Grade 4, <1.5. Hyperkalemia (mmol/L), Grade 3, >6.0-7.0; Grade 4, >7.0. Hypokalemia (mmol/L), Grade 3, <3.0-2.5; Grade 4, <2.5. Hypernatremia (mmol/L), Grade 3, >155-160; Grade 4, >160. Hyponatremia (mmol/L), Grade 3, <130-120; Grade 4, <120. Phosphorus (mmol/L), Grade 3, <0.6-0.3; Grade 4, <0.3. Prothrombin time (seconds), Grade 3, >2.0; Grade 4, not defined.
Time Frame: From Day 2 of Cycle 1 to up to 30 days after last dose of study drug (up to approximately 49 months)
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Dasatinib, 50 mg + Docetaxel, 60 mg/m^2 | Dasatinib, 50 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 70 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 120 mg + Docetaxel, 75 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 34 | 3
Participants
  Absolute neutrophil count | 0 | 0 | 0 | 1 | 0
  Hemoglobin | 0 | 0 | 0 | 0 | 0
  Platelet count | 0 | 0 | 0 | 0 | 0
  Leukocytes | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase (ALT) | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase (AST) | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase (ALP) | 1 | 1 | 0 | 1 | 0
  Total bilirubin | 0 | 0 | 0 | 0 | 0
  Hypercalcemia | 0 | 0 | 0 | 0 | 0
  Hypocalcemia | 0 | 0 | 0 | 1 | 0
  Creatinine | 0 | 0 | 0 | 0 | 0
  Hyperkalemia | 0 | 0 | 0 | 1 | 0
  Hypokalemia | 0 | 0 | 0 | 0 | 1
  Hypernatremia | 0 | 0 | 0 | 0 | 0
  Hyponatremia | 0 | 0 | 0 | 2 | 0
  Phosphorus, inorganic | 0 | 1 | 0 | 1 | 0
  Prothrombin time | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From 1st dose, Day 1 to up to 30 days after last dose of study drug (approximately 49 months + 30 days)
Arm/Group | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 120 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 50 mg + Docetaxel, 60 mg/m^2 | Dasatinib, 50 mg + Docetaxel, 75 mg/m^2 | Dasatinib, 70 mg + Docetaxel, 75 mg/m^2
Serious Adverse Events (participants affected / at risk) | 14/34 | 1/3 | 1/3 | 0/3 | 1/3
Other Adverse Events (participants affected / at risk) | 34/34 | 3/3 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2 (N=34) | Dasatinib, 120 mg + Docetaxel, 75 mg/m^2 (N=3) | Dasatinib, 50 mg + Docetaxel, 60 mg/m^2 (N=3) | Dasatinib, 50 mg + Docetaxel, 75 mg/m^2 (N=3) | Dasatinib, 70 mg + Docetaxel, 75 mg/m^2 (N=3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 100 mg + Docetaxel, 75 mg/m^2 (N=34) | Dasatinib, 120 mg + Docetaxel, 75 mg/m^2 (N=3) | Dasatinib, 50 mg + Docetaxel, 60 mg/m^2 (N=3) | Dasatinib, 50 mg + Docetaxel, 75 mg/m^2 (N=3) | Dasatinib, 70 mg + Docetaxel, 75 mg/m^2 (N=3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0
Pain (General disorders) | 6 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 4 | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 9 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 2 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 6 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 8 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 5 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 2 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 2 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 1 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 6 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 4 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 6 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 6 | 0 | 1 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 9 | 2 | 2 | 1 | 0
Dysgeusia (Nervous system disorders) | 17 | 2 | 2 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 27 | 1 | 3 | 1 | 3
Laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 6 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 2 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Urethral pain (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 5 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 5 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Oedema (General disorders) | 2 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 17 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 2 | 1 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 3 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 4 | 0 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 20 | 0 | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 10 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 4 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 2 | 1 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time shortened (Investigations) | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 25 | 1 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 3 | 0 | 0 | 0 | 0
Chills (General disorders) | 2 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 25 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 2 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 14 | 1 | 1 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.